CLINICAL TRIAL: NCT01995149
Title: Effect of Weight Loss on Lipids Concentration and Cholesterol Metabolism in Overweight and Obese Subjects With Primary Hypercholesterolemia.
Brief Title: Effect of Weight Loss on Cholesterol Metabolism in Hereditary Hypercholesterolemias and Overweight or Obesity.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto Aragones de Ciencias de la Salud (Other Government)
Collaborators: Hospital Clinic of Barcelona (Other); Instituto de Salud Carlos III (Other Government)
Responsible Party: Principal Investigator, Fernando Civeira, Professor, Instituto Aragones de Ciencias de la Salud
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: I+CS;CEICA-B80; I+CS-HUMS-B80 (Other: I+CS/HUMS-B80)
Record Dates: First submitted 2013-11-21; First posted 2013-11-26 (Estimated); Last update posted 2013-11-26 (Estimated); Status verified 2013-11

CONDITIONS: Familial Hypercholesterolemias; Weight Loss; Familial Combined Hypercholesterolemia; Obesity
Keywords: Familial Hypercholesterolemia; Familial Combined Hypercholesterolemia; Weight loss; Lipids; Phytosterols; Obesity; Overweight.; Lipids
MeSH Terms: conditions — Hyperlipoproteinemia Type II; Weight Loss; Obesity; Overweight | interventions — Diet Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Weight loss and dietary intervention (Experimental): The weight loss intervention had a total duration of 6 months. Each participant's caloric prescription represented a deficit of 600 kcal per day as calculated from the person's resting energy expenditure and activity level using the Harris-Benedict equation. In general, prescribed energy intake was between 1200 kcal and 1600 kcal/day. Dietary composition consisted on 50-55% of carbohydrates, 15-20% of protein and 30% of fat and included a wide variety of foods typical of a Mediterranean diet. Patients were also provided with recipes and shopping counselling to improve intervention compliance and to achieve the weight loss goal. Individual consultations with a nutritionist were performed twice a month to motivate the weight loss and reinforce the intervention.
  Interventions: Behavioral: Weight loss and dietary intervention

INTERVENTIONS:
Behavioral: Weight loss and dietary intervention — The weight loss intervention had a total duration of 6 months. Each participant's caloric prescription represented a deficit of 600 kcal per day as calculated from the person's resting energy expenditure and activity level using the Harris-Benedict equation. In general, prescribed energy intake was between 1200 kcal and 1600 kcal/day. Dietary composition consisted on 50-55% of carbohydrates, 15-20% of protein and 30% of fat and included a wide variety of foods typical of a Mediterranean diet. Patients were also provided with recipes and shopping counselling to improve intervention compliance and to achieve the weight loss goal. Individual consultations with a nutritionist were performed twice a month to motivate the weight loss and reinforce the intervention.

SUMMARY:
Background: Lipid lowering response to weight loss in subjects with genetic hyperlipidemias and overweight or obesity and its effect on cholesterol metabolism has not been studied.

Objective: To explore the effects of weight loss on lipid values and cholesterol metabolism, by measuring circulating non-cholesterol sterols, in overweight or obese subjects with genetic hypercholesterolemias.

Design: The investigators conducted a 6-months weight loss intervention in subjects with the diagnosis of familial hypercholesterolemia (FH) or familial combined hyperlipidemia (FCHL), body mass index >25 kg/m2, steady weight (±3 kg in the last 3 months) and absence of lipid lowering drugs in the previous 5 weeks. They were advised to follow a hypocaloric diet with a deficit of 600 kcal (30% fat, 15% protein, and 55% carbohydrates) per day as calculated from the person's resting energy expenditure and activity level. Anthropometric data, biochemical analysis including lipids, apolipoproteins and non-cholesterol sterols were evaluated at baseline, 3 months and 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years.
* Diagnosis of Familial Combined Hyperlipidemia* and Familial Hypercholesterolemia**.
* Body mass index > 25 kg/m2.
* Steady weight (±3 kg in the last 3 months).
* Absence of lipid lowering drugs including sterols supplements in the previous 5 weeks.

  * Familial Combined Hyperlipidemia diagnosis was based on the presence of primary combined hyperlipidaemia in untreated patients whose serum cholesterol and triglyceride concentrations were above the sex- and age-specific 90th percentiles for the Spanish population, serum total apolipoprotein B concentration ≥ 120 mg/dL and there was at least one first-degree relative with hyperlipidemia (total cholesterol and/or triglycerides >90th percentile) (Gómez-Gerique JA et al; 1999).

    * Familial Hypercholesterolemia was diagnosed in subjects with off-treatment LDL cholesterol concentrations above the age- and sex-specific 95th percentile of a Spanish reference population, triglyceride below 200 mg/dL and familial vertical transmission with at least one first-degree relative with LDL cholesterol above age- and sex-specific 95th percentiles (Gómez-Gerique JA et al; 1999).

Exclusion Criteria:

* Alcohol consumption >30 gr/day.
* Uncontrolled type-2 diabetes (HbA1c >8%).
* Any other disease that could interfere with the ability to comply with the study protocol were excluded
* Personal history of cardiovascular disease, very high risk as defined by the presence of ≥ 2 major risk factors, or total cholesterol ≥ 350 mg/dL since lipid-lowering drug were considered highly recommended.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2010-06; Primary Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Change in lipids and non-cholesterol sterols concentration | After 6 months of intervention
  Main outcome it the variation of:
  * Lipids: Total cholesterol, LDL cholesterol, HDL cholesterol, tryglicerides and apolipoprotein B.
  * Non-cholesterol sterols: Phytosterols (campesterol, stigmasterol and sitosterols) and cholestanol (which are stated as subrogate markers of intestinal cholesterol absorption) and desmosterol, lathosterol and lanosterol (cholesterol synthesis markers).

CONTACTS AND LOCATIONS:
Overall Officials: Fernando Civeira, MD, PhD, Principal Investigator — Unidad de Lípidos/Laboratorio de Investigación Molecular; Hospital Universitario Miguel Servet; Instituto Aragonés de Ciencias de la Salud

REFERENCES:
- [Derived] Mateo-Gallego R, Perez-Calahorra S, Cofan M, Baila-Rueda L, Cenarro A, Ros E, Puzo J, Civeira F. Serum lipid responses to weight loss differ between overweight adults with familial hypercholesterolemia and those with familial combined hyperlipidemia. J Nutr. 2014 Aug;144(8):1219-26. doi: 10.3945/jn.114.191775. Epub 2014 Jun 4. PMID 24899155